CLINICAL TRIAL: NCT02313051
Title: A Multicenter, Randomized Phase ll Study of Letrozole Versus Letrozole Plus Everolimus for Hormone Receptor-PositivePremenopausal Women With Recurrent or Metastatic Breast Cancer on Goserelin Treatment After Progression on Tamoxifen
Brief Title: Everolimus trIal for Advanced prememopausaL Breast Cancer Patients
Acronym: MIRACLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Binghe Xu, Director of department of medical oncology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBCSG016
Record Dates: First submitted 2014-11-24; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-11

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer, everolimus
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Goserelin; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus arm (Experimental): Everolimus+letrozole
  Interventions: Drug: Everolimus; Drug: Goserelin; Drug: Letrozole
- Controll arm (Active Comparator): letrozole alone, and when progress, followed by everolimus
  Interventions: Drug: Goserelin; Drug: Letrozole

INTERVENTIONS:
Drug: Everolimus — mTOR inhibitor
  Other Names: Certican; Rad001
  Arms: Everolimus arm
Drug: Goserelin
  Other Names: Zoladex
Drug: Letrozole
  Other Names: Femara

SUMMARY:
Everolimus has been approved to be effective when used with exemestane after progression on non-steroidal aromatase inhibitors in postmenopausal women based on the BOLERO-2 clinical trial. However, the superiority of addition of everolimus to endocrine therapy hasn't been established in the premenopausal women. This is a phase 2, multicentre clinical trial to evaluate the role of everolimus in the first-line endocrine treatment of premenopausal MBC patients after progression on tamoxifen.

DETAILED DESCRIPTION:
Endocrine therapy is the cornerstone of treatment for patients with hormone receptor (HR)-positive advanced breast cancer. The selection of endocrine agents takes account of the menopausal status, the type of previous adjuvant endocrine treatment, the disease free interval and past medical history.

In premenopausal women with HR-positive advanced breast cancer, ovarian function suppression combined with aromatase inhibitors is a standard first-line choice of hormone treatment, especially patients progressed after tamoxifen. Unfortunately, not all patients have a response to first-line endocrine therapy, and even patients who have a response will eventually become resistant.

An emerging mechanism of endocrine resistance in aberrant signaling through the phosphatidylinositol 3-kinase (PI3K)-Akt-mammalian target of rapamycin (mTOR) signaling pathway7-9. Growing evidence supports a close interaction between the mTOR pathway and ER signaling. Everolimus is a sirolimus derivative that inhibits mTORactivation11. In preclinical models, the use of everolimus in combination with aromatase inhibitors results in synergistic inhibition of the proliferation and induction of apoptosis12. In a randomized, phase 2 study comparing neoadjuvant everolimus plus letrozole with letrozole alone in patients with newly diagnosed ER-positive breast cancer, the response rate for the combination was higher than that for letrozole alone. Recently, the Breast Cancer Trials of Oral Everolimus-2 (BOLERO-2) study showed that the addition of everolimus to exemestane significantly improved progression-free survival, with observed medians of 11 and 4 months, corresponding to a 62% reduction in the hazard ratio14 which is impressive and practice changing.

However, different from western countries, the majority (50-55%) of patients are premenopausal women in Asia including China.The benefit of everolimus plus endocrine therapy in premenopausal women have not yet been well delineated. Although there was a report that efficacy was comparable between premenopausal metastatic breast cancer patients treated with letrozole plus goserelin and postmenopausal patients treated with letrozole alone as first line hormone therapy, it is generally accepted that endocrine treatment outcome in premenopausal women, especially in younger age is known to be poor. So the addition of everolimusin this population would be a potential viable treatment option to overcome resistance to endocrine therapies that needs to be evaluated.

In addition, the feasibility of patients progressed on the endocrine continue to receive the same endocrine agent plus everolimus is unclear. At the same time, the difference between concurrent and sequential medication of endocrine agent and everolimus is not yet addressed.

Based on this rationale, the investigators introduced randomized trial to evaluate the efficacy of addition of everolimus to letrozole with LHRH agonist in premenopausal metastatic breast cancer patients who failed to tamoxifen treatment and also explore the best schedule of endocrine therapy together with everolimus.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 years of age) with metastatic or locally advanced breast cancer not amenable to curative surgery.
* Histological confirmation of estrogen and/or progesterone-receptor positive (ER+), human epidermal growth factor receptor 2 negative (HER2 -) breast cancer.

ER/PR positive: nuclear reaction > 1%, HER2 negative: HER2; IHC 0,1+ or FISH/CISH (-) in case of IHC 2+

* Patients who:

  * received Tamoxifen for at least 6 months during adjuvant treatment and recurred during or within 24 months after the end of adjuvant treatment completion,
  * progressed during tamoxifen treatment for advanced disease.
* Pre-menopausal status was defined as either :
* The patient has a history of regular menstrual periods within 12 weeks prior to study enrollment
* The patient has FSH and E2 levels with in pre-menopausal range based on local laboratory assessments measured (i.e, FSH ≤ 40 mIU/mL and E2 ≥10 pg/mL)within 12 weeks prior to study enrollment.
* ECOG performance status of 0,1, or 2
* At least one measurable lesion or mainly lytic bone lesions in the absence of measurable disease(RECIST1.1)
* Adequate bone marrow, hepatic, and renal function
* Adequate bone marrow and coagulation function as shown by:
* Absolute neutrophil count (ANC) ≥ 1.5 109/L;Platelets>100 x109/L;Hemoglobin (Hgb) > 9.0g/dLINR < 2
* Adequate liver function as shown by:
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5x ULN (or <5 if hepatic metastases are present)
* Total serum bilirubin < 1.5 x ULN (<3 x ULN for patients known to have Gilberts Syndrome)
* Adequate renal function as shown by:
* Serum creatinine< 1.5 x ULN
* Fasting serum cholesterol <300 mg/dL or 7.75 mmol/L and fasting triglycerides <2.5 x ULN. In case one or both of these thresholds are exceeded, the patient can only be included after initiation of statin therapy and when the above mentioned values have been achieved.
* Written informed consent

Exclusion Criteria:

* Patients who have received endocrine treatment other than Tamoxifen for adjuvant or metastatic/locally advanced breast cancer.
* Patients who have received goserelin at adjuvant setting
* Patients who received more than one line of chemotherapy for metastatic or locally advanced breast cancer
* Previous treatment with mTOR inhibitors.
* Another malignancy within 5 years prior to enrollment with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer.
* Symptomatic brain or other CNS metastases
* Patients receiving chronic treatment with immunosuppressive agents.
* Any severe and/or uncontrolled medical conditions, eg. currently active infection
* Pregnant or lactating
* Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 6 months after last patient was evaluated
  the time from randomization to the time of disease progression or relapse or death

SECONDARY OUTCOMES:
Overall survival | 1 year after the last patient was followed-up
  time from randomization to death
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | during screening and treatment, withing 28 days after last medication
Clinical benefit rate | at the time of tumor assessment of last patient
Duration of clinical benefit | 6 months after last patient was evaluated
  from the date of confirmed response to the confirmed progression

CONTACTS AND LOCATIONS:
Overall Officials: Bing he Xu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Fan Y, Sun T, Shao Z, Zhang Q, Ouyang Q, Tong Z, Wang S, Luo Y, Teng Y, Wang X, Wang S, Liu Q, Feng J, Shen K, Song Y, Wang J, Ma F, Li Q, Zhang P, Xu B. Effectiveness of Adding Everolimus to the First-line Treatment of Advanced Breast Cancer in Premenopausal Women Who Experienced Disease Progression While Receiving Selective Estrogen Receptor Modulators: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):e213428. doi: 10.1001/jamaoncol.2021.3428. Epub 2021 Oct 21. PMID 34436536